CLINICAL TRIAL: NCT02531607
Title: Lipidomics, Proteomics, Micro RNAs and Volatile Organic Compounds Biomarkers in Bile and Serum in the Diagnosis of Malignant Biliary Strictures
Brief Title: Lipidomics, Proteomics, Micro RNAs and Volatile Organic Compounds (VOC)
Status: Active, not recruiting | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 649074
Record Dates: First submitted 2015-02-11; First posted 2015-08-24 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bile and blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood and bile — 20ml of blood will be obtained from consented participants. 5ml of bile will be collected during the endoscopic procedure.

SUMMARY:
This is a non-randomized natural history protocol in which patients undergoing surgery or endoscopy for suspected/ diagnosed pancreaticobiliary strictures are assigned to a) control (chronic pancreatitis, no pancreatic neoplasm, primary sclerosing cholangitis), b) non-carcinoma (bile duct stones, papillary stenosis, ), c) carcinoma non-pancreatic (ampullary and distal bile duct or cholangiocarcinoma) and d) pancreatic ductal adenocarcinoma (pancreatic cancer.

DETAILED DESCRIPTION:
Visit 1 for all participants will consist of going over the Informed Consent form and talking with the patient about the study. If the patient agrees to participate, he/she will be asked to sign the form, and a copy will be given to him/her for his/her records. This will be conducted during the day of the endoscopic procedure before the participant is under anesthesia.

Consented participants will have 20ml of blood collected via venipuncture of peripheral vein drawn by the endoscopy unit staff during their endoscopy procedure. The blood will be collected into heparinized vacutainers and immediately labeled with study specific code identifier and placed at 4⁰C until processed (within 24hr).

For clinical purposes, tissue may be removed during the endoscopic procedures. This tissue will be given to the Diagnostic Pathology (DP) personnel associated with the case for analysis. The diagnostic sample will be processed for DP use and stored in the DP active archives. No additional tissue will be taken solely for the purposes of this research study. However, if DP approves the use of the remaining clinical diagnostic, small cores or slides will be taken after the diagnostic use from the approved paraffin-embedded tissue blocks for use in comparison/confirmatory analyses to the bile and blood analyses done for this research project.

During the endoscopic procedures a 5ml aspiration of bile fluid will be collected for this study with the endoscopic instrument. The fluid will be transferred to a sterile tube, sealed, and placed at 4⁰C until processed (within 24hr). Both blood and fluids samples will be transferred to Translational Research Institute (TRI) R&D for analysis.

Follow Up (follow up will take place for all groups listed on page 7 of the protocol under "Study Design" with the exception of group B) 2 weeks post procedure- A member of the research staff will call the participant to assess for any complications Periodic medical record auditing for outcome data will be collected every three months for up to 1 year after enrollment.

One year post procedure- A member of the research staff will call the participant to assess for any complications

ELIGIBILITY:
Inclusion Criteria:

Screening Criteria for Potential Participants in the Study

1. Age: ≥18years old
2. Treatment: scheduled for clinical reason to undergo an ERCP at the CIE
3. Suspected of having biliary or pancreatic disease other than cancer (chronic pancreatitis, benign biliary strictures, post-liver transplant strictures, common bile duct stones, sphincter of Oddi dysfunction or suspected of having pancreatic or peri-ampullary malignancy (including pancreatic ductal adenocarcinoma, distal cholangiocarcinoma, ampullary carcinoma, duodenal, carcinoma
4. Clinical or image data suggestive of pancreatic disease or the need for gastrointestinal or pancreatic inspection.
5. Willing and mentally able to provide consent

Exclusion Criteria:

1. Age: <18years old
2. Pregnant women
3. Post-bariatric surgery, hepaticojejunostomy and Bilroth II patients undergoing ERCP.
4. Not scheduled for endoscopic procedures for clinical reasons
5. No clinical or image data suggestive of need for clinical intervention (Endoscopy)
6. Not willing or able to sign informed consent..

Ages: 19 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for ERCP at the Center for Interventional Endoscopy (CIE)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-11-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of biomarkers in the diagnosis of cancer | one year
  Comparative efficacy of biomarkers, brush cytology, fluorescence in situ hybridization (FISH), carbohydrate antigen 19-9 (CA 19-9) and biliary and blood biomarkers (lipidomics, proteomics, micro RNAs and VOCs) in the diagnosis of malignancy.

SECONDARY OUTCOMES:
Medical Record Review | one year
  Subjects who do not have a differential diagnosis of either cancer, biliary or pancreatic disease at the time of the index Endoscopic retrograde cholangiopancreatography (ERCP) will have their medical record reviewed quarterly for new diagnoses or procedures related to pancreatic malignancy, peri-ampullary malignancy, biliary disease, or pancreatic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pratley, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Navaneethan U, Spencer C, Zhu X, Vargo JJ, Grove D, Dweik RA. Volatile organic compounds in bile can distinguish pancreatic cancer from chronic pancreatitis: a prospective observational study. Endoscopy. 2021 Jul;53(7):732-736. doi: 10.1055/a-1255-9169. Epub 2020 Sep 4. PMID 32894868